CLINICAL TRIAL: NCT00379405
Title: Open-label, Comparative and Randomised Pilot Study to Evaluate the Efficacy and Safety of Saquinavir/Ritonavir in Single Therapy vs Standard HAART Therapy as Maintenance Therapy.
Brief Title: Saquinavir/Ritonavir in Single Therapy as Maintenance Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQV/RTV-MONOTERAPIA; 2006-001136-47
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Saquinavir/ritonavir; Single therapy; Virological efficacy; Safety; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Saquinavir (Invirase): 2 capsules (500 mg) / 12 hours
  Interventions: Drug: Saquinavir/Ritonavir : 2 capsules (500 mg) / 12 hours
- 2 (No Intervention): IP o NNUCS + 2 NUCS as a HAART therapy .

INTERVENTIONS:
Drug: Saquinavir/Ritonavir : 2 capsules (500 mg) / 12 hours — Saquinavir/Ritonavir: 2 capsules (500 mg) / 12 hours
  Other Names: Invirase
  Arms: A

SUMMARY:
Study the efficacy of Saquinavir/Ritonavir when given in single therapy as maintenance therapy, compared to standard HAART therapies.

DETAILED DESCRIPTION:
Different therapeutic strategies have been investigated to improve adherence to treatment and reduce toxicity. Both the reduction in the number of doses and the number of daily tablets have led to an improvement in therapeutic compliance. Similarly, the administration of new treatment regimens with a reduced number of tablets a day and without NTRI may be clinically useful in improving compliance with HAART and limiting NTRI-associated toxicity. These would comprise combinations of a PI, boosted with ritonavir, plus a non-Nucleoside and single therapy with PIs boosted with ritonavir.

In this regard, the results obtained with lopinavir/ritonavir and with atazanavir/ritonavir are very promising and open up a possible channel of research with other PIs boosted with low doses of ritonavir.

There are other PIs whose antiretroviral efficacy has also been demonstrated, such as saquinavir, but whose economic cost is much lower. Furthermore, saquinavir has a low toxicity profile, and the availability of saquinavir 500 mg facilitates comfortable administration, since it makes it possible to reduce the number of daily tablets to more than half.

Moreover, it is important to take into account that the incidence of mutations that confer resistance to saquinavir on patients that fail on combinations including this PI is very low, which makes it possible to reuse the drug in future treatment regimens or salvage patients with other PI All these characteristics (high intrinsic potency, low number of tablets, low toxicity, low potential of selection of resistant viral strains in combination with ritonavir, and low economic cost) make single therapy with the new formulation of saquinavir, boosted with low doses of ritonavir, a possible therapeutic option as maintenance strategy in HIV-infected patients with maintained suppression of the viral load.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by HIV-1 (at least one documented positive Western-Blot).
* Age > 18 years.
* Patients on antiretroviral treatment (standard HAART therapy) for at least six months.
* HIV-1 plasma viral load <50 copies/mL (documented in at least two determinations performed over the six months prior to the inclusion visit).
* Patients without evidence of previous virological failure to IP
* Absence of opportunistic infections and/or tumours in the three months prior to inclusion.
* Subject able to follow the treatment period, without any suspicion of poor adherence during previous antiretroviral treatments.
* Signature of the informed consent.

Exclusion Criteria:

* Suspicion of unsuitable antiretroviral treatment compliance.
* Documented existence of any of the primary mutations in the protease gene or 3 or more of the following: L10F/I/R/V, K20M/R, M36I/V, I54L/T/V, L63P, A71T/V , V82A/F/T/S, I84A/V OR L90M.
* Known allergic hypersensitivity to any of the investigational drugs or any similar drug.
* Hepatic tests (AST, ALT, GGT) > or equal to 5 times the upper limit of normality during the three months prior to the screening visit
* Presence of renal impairment (creatinine > or equal to 1.5 times the upper limit of normality).
* Pregnancy or breastfeeding. Refusal to use reliable contraceptive methods during the study period.
* Participation in another clinical trial wich entail the antiretroviral treatment modification.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Virological response: Viral Load | weeks 24 and 48

SECONDARY OUTCOMES:
CD4 and CD8 lymphocyte count. | weeks 24 and 48
Physical Exploration: including weight, height, index waist/hip (the abdominal perimeter is measured between the last floating rib and the iliac crest), assessment of changes in body fat distribution,... | weeks 24 and 48
Karnofsky Index. | weeks 24 and 48
Adverse events. | during the 48 weeks of follow-up
Trough plasma concentrations of Saquinavir. | during the 48 weeks of follow-up
Lipid study in plasma (total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides) | during the 48 weeks of follow-up
Serology for Hepatitis B and C virus. | at baseline visit
Assessment of treatment adherence. | at baseline and weeks 4, 12, 24, 36 and 48
Assessment of quality of life (by means of the MOS-HIV questionnaire). | at baseline and weeks 4, 12, 24, 36 and 48
Genotype if virological failure. | at any time of study if it is necessary

CONTACTS AND LOCATIONS:
Overall Officials: Clotet Bonaventura, MD,PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol. Badalona (Barcelona); Negredo Eugenia, MD,PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol. Badalona. (Barcelona); Echeverria Patricia, MD,PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol. Badalona. (Barcelona); Molto Jose, MD,PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol. Badalona. (Barcelona); Pere Domingo, MD, PhD, Principal Investigator — Hospital de Sant Pau
Locations (2):
- Spain (2):
  - Germans Trias i Pujol University Hospital, Badalona, Barcelona
  - Hospital del Sant Pau., Barcelona